CLINICAL TRIAL: NCT07187648
Title: The Effect of Golden Rice Cookies With Piper Crocatum on Fasting Blood Sugar and Quality of Life in People Living With HIV With Hyperglycemia
Brief Title: Golden Rice Cookies With Piper Crocatum for Blood Glucose Control and Quality of Life in People Living With HIV With Hyperglycemia
Acronym: GRC-HIV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Deni Wardani, Principal Investigator, Hasanuddin University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UH2506067
Record Dates: First submitted 2025-09-07; First posted 2025-09-23 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections; Nutritional Intervention; Blood Glucose; Quality of Life
Keywords: HIV; Golden Rice; Quality of Life; Blood Glucose
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in parallel to one of two groups: the intervention group receiving Golden Rice Cookies with Piper crocatum or the control group receiving placebo. Both groups will consume their assigned cookies daily for 28 days
Who Masked: Participant
Masking Description: Only participants are blinded to group assignment. The intervention and control cookies are made to appear similar in packaging and portion, so participants do not know whether they are receiving Golden Rice Cookies with Piper crocatum or control cookies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Golden Rice Cookies With Piper crocatum (Experimental): Participants in this group will consume Golden Rice cookies enriched with Piper crocatum. Each participant will receive 20 g twice daily (40 g/day total) for 28 days. The cookies are designed to be iso-caloric with the control cookies and packaged identically to maintain participant blinding.
  Interventions: Dietary Supplement: Golden Rice Cookies With Piper crocatum
- so-Caloric Cookies Without Golden Rice and Piper crocatum (Placebo Comparator): Participants in this group will consume placebo cookies made from standard flour without Golden Rice and without Piper crocatum. Each participant will receive 20 g twice daily (40 g/day total) for 28 days. The cookies are calorie-matched and designed to resemble the intervention cookies in appearance but do not contain the active ingredients.
  Interventions: Other: Iso-Caloric Control Cookies (Placebo)

INTERVENTIONS:
Dietary Supplement: Golden Rice Cookies With Piper crocatum — Golden Rice cookies enriched with Piper crocatum were formulated as a functional food containing β-carotene and bioactive compounds (polyphenols, flavonoids, tannins). Participants in the experimental arm consume 20 g twice daily (40 g/day total) for 28 days. The cookies are iso-caloric with control cookies but differ by inclusion of Golden Rice and Piper crocatum.
  Arms: Golden Rice Cookies With Piper crocatum
Other: Iso-Caloric Control Cookies (Placebo) — Iso-caloric cookies made from standard flour without Golden Rice and without Piper crocatum. Participants in the control arm consume 20 g twice daily (40 g/day total) for 28 days. The cookies are designed to match the intervention cookies in calories and appearance but do not contain the active ingredients.
  Arms: so-Caloric Cookies Without Golden Rice and Piper crocatum

SUMMARY:
The goal of this clinical trial is to learn if Golden Rice Cookies with Piper crocatum can help improve fasting blood sugar and quality of life in people living with HIV who have hyperglycemia (GRC-HIV). It will also learn about the safety and acceptability of this dietary intervention.

The main questions it aims to answer are:

Does Golden Rice Cookies with Piper crocatum lower fasting blood sugar levels in PLHIV with hyperglycemia? Does Golden Rice Cookies with Piper crocatum improve quality of life in PLHIV with hyperglycemia? Researchers will compare Golden Rice Cookies with Piper crocatum to control cookies (iso-caloric cookies without Golden Rice and Piper crocatum) to see if Golden Rice Cookies are effective.

Participants will:

Consume either Golden Rice Cookies with Piper crocatum or control cookies every day for 28 days Visit the clinic at baseline and follow-up for checkups, laboratory tests, and questionnaires Record their daily cookie consumption and any symptoms or side effects in a diary

DETAILED DESCRIPTION:
People living with HIV (PLHIV) are at higher risk of developing hyperglycemia due to long-term antiretroviral therapy (ART), metabolic complications, and lifestyle factors. Hyperglycemia not only worsens the prognosis of HIV but also negatively affects quality of life. Dietary interventions using functional foods may provide a safe and acceptable strategy to address this issue.

Golden Rice is biofortified with β-carotene, which has been associated with improved insulin sensitivity and reduced glycemic response. Piper crocatum (red betel leaf) contains polyphenols, flavonoids, and tannins with antidiabetic, antioxidant, and anti-inflammatory properties. Combining Golden Rice and Piper crocatum in a practical cookie form offers a potentially effective and acceptable intervention for PLHIV with hyperglycemia.

This trial is designed to evaluate whether daily consumption of Golden Rice Cookies enriched with Piper crocatum can improve fasting plasma glucose and health-related quality of life in PLHIV with hyperglycemia compared to iso-caloric control cookies. The findings may contribute to evidence-based dietary strategies to improve metabolic outcomes and well-being in PLHIV.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive diagnosis based on medically documented serological test results (ELISA/Western Blot/rapid test).
* Age 35-59 years.
* Suffering from hyperglycemia, defined by a Fasting Blood Sugar (FBS) value of ≥ 100 mg/dl (prediabetes or diabetes), according to ADA (American Diabetes Association) standards and a physician's report.
* Taking antiretroviral therapy (ART) for at least the past 2 years to ensure stable clinical status.
* CD4 count ≥ 200 cells/mm³, to exclude participants with severely compromised immunity that could impact metabolism and quality of life.
* Not currently undergoing strict diet therapy or other nutritional interventions to avoid nutritional bias.
* Willing to sign informed consent and participate in all stages of the study

Exclusion Criteria:

* Having acute complications of HIV/AIDS, such as severe opportunistic infections, that may interfere with interventions or quality of life measurements.
* Having a history of other chronic diseases that affect glucose metabolism, such as advanced chronic kidney disease, active cancer, hyperthyroidism, or severe liver disease.
* Using medications that can affect blood sugar levels (e.g., steroids, thiazide diuretics, or other hyperglycemic drugs) in the past month.
* Allergies to ingredients in Golden Rice Cookies (Red Rice) or Piper crocatum.
* Being pregnant or breastfeeding.
* Participating in other nutrition intervention programs, intensive physical training.
* Inability to read or understand instructions (e.g., due to severe cognitive impairment) that may interfere with completing the quality of life questionnaire.

Ages: 35 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Fasting Plasma Glucose | Baseline and 28 days
  Change in fasting plasma glucose level from baseline to Day 28, measured using enzymatic method after 8-10 hours of fasting. Measurement scale:
  1. <100 mg/dL = Normal
  2. 100-125 mg/dL = Prediabetes
  3. ≥126 mg/dL = Diabetes Mellitus
Change in Health-Related Quality of Life | Baseline and 28 days
  Change in quality of life score assessed using WHOQOL-HIV BREF questionnaire from baseline to Day 28.
  Measurement results:
  1. Low Quality of Life: <41
  2. Moderate Quality of Life: 41-60
  3. High Quality of Life ≥60

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because of confidentiality and privacy considerations for people living with HIV, as well as institutional data protection policies.

REFERENCES:
- [Result] Tang G, Qin J, Dolnikowski GG, Russell RM, Grusak MA. Golden Rice is an effective source of vitamin A. Am J Clin Nutr. 2009 Jun;89(6):1776-83. doi: 10.3945/ajcn.2008.27119. Epub 2009 Apr 15. PMID 19369372
- [Result] Setyawati A, Wahyuningsih MSH, Nugrahaningsih DAA, Effendy C, Fneish F, Fortwengel G. Piper crocatum Ruiz & Pav. ameliorates wound healing through p53, E-cadherin and SOD1 pathways on wounded hyperglycemia fibroblasts. Saudi J Biol Sci. 2021 Dec;28(12):7257-7268. doi: 10.1016/j.sjbs.2021.08.039. Epub 2021 Aug 19. PMID 34867030
- [Result] Zuniga JA, Jang DE, Walker G, Ohueri CW, A Garcia A. Differences in Health-Related Quality of Life Predictors in People Living With HIV With and Without Diabetes. J Assoc Nurses AIDS Care. 2020 Sep-Oct;31(5):544-552. doi: 10.1097/JNC.0000000000000138. PMID 31789685
- See also: Official website of the Faculty of Nursing, Universitas Hasanuddin provides information on academic programs (including Master of Nursing ), research activities, organizational structure, and institutional collaborations. — https://nursing.unhas.ac.id/